CLINICAL TRIAL: NCT01345045
Title: A Multicenter, Randomized, Double-Blind, Placebo and Active Controlled Study Comparing the Analgesic Efficacy and Safety of ABT-639 to Placebo in Subjects With Diabetic Neuropathic Pain
Brief Title: A Multicenter Study Comparing the Analgesic Effects and Safety of ABT-639 Compared to Placebo in Subjects With Diabetic Neuropathic Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M11-891; 2010-024359-99 (EudraCT Number)
Record Dates: First submitted 2011-04-28; First posted 2011-04-29 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Diabetic Neuropathic Pain
Keywords: Diabetic Asymmetric Polyneuropathy; Symmetric Diabetic Proximal Motor Neuropathy; Diabetic Mononeuropathy Simplex,; Diabetic Autonomic Neuropathy,; Diabetic Amyotrophy; Mononeuropathy; Diabetic Neuropathy; Asymmetric Diabetic Proximal Motor Neuropathy; Diabetic Polyneuropathy; Painful; Diabetic Mononeuropathy; Neuralgia
MeSH Terms: conditions — Diabetic Neuropathies; Mononeuropathies; Pain; Neuralgia | interventions — 4-chloro-2-fluoro-N-(2-fluorophenyl)-5-(hexahydropyrrolo(1,2-a)pyrazin-2(1H)-ylcarbonyl)benzenesulfonamide; Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- ABT-639 (Experimental): ABT-639 twice daily for 6 weeks
  Interventions: Drug: ABT-639
- pregabalin (Active Comparator): pregabalin starting dose twice daily for week one then titrated up to maintenance dose twice daily for duration of the study
  Interventions: Drug: pregabalin
- Placebo (Placebo Comparator): Placebo twice daily for 6 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ABT-639 — ABT-639 Twice Daily for six weeks.
  Arms: ABT-639
Drug: pregabalin — pregabalin starting dose twice daily for 1 week then titrated to maintenance dose twice daily for the remainder of the study.
  Other Names: Lyrica
  Arms: pregabalin
Drug: Placebo — Placebo twice daily for 6 weeks.
  Arms: Placebo

SUMMARY:
People with diabetes can, over time develop nerve damage throughout the body with symptoms such as pain, tingling, or numbness (loss of feeling) in the hands, arms, feet and legs.

ELIGIBILITY:
Inclusion Criteria:

* Subject is between the ages of 18 to 75 years with a diagnosis of diabetes mellitus and must have a diagnosis of painful distal symmetric diabetic polyneuropathy and presence of ongoing pain due to diabetic peripheral neuropathy for at least 6 months.
* Subject must have an average score of greater than or equal to ( ≥) 4 on the 24 hour average pain score (0-10 numerical rating scale) collected over approximately 7 days prior to the Baseline Visit.

Exclusion Criteria:

* Subject has clinically symptomatic neuropathic pain conditions that can not be distinguished from Diabetic Neuropathic Pain (DNP) or interfere with the pain assessments of DNP.
* A subject has newly diagnosed or clinically significant medical conditions or mental disorders that would preclude participation or would interfere with DNP assessments or other functions.
* Subject has clinically significant abnormalities in clinical laboratory tests.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2011-04; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
A mean of 24-hour average pain score measured by an 11-point Numeric Rating Scale (NRS) based on subject's daily diary | Weekly started at Baseline, Week 1, Week 2, Week 4, and Week 6 (End of Study)
  Daily questions asked on a hand held diary

SECONDARY OUTCOMES:
Patient's Global Impression of Change | Week 2, Week 4 and Week 6 (End of Study)
  Paper questionnaire
Brief Pain Inventory (BPI) (short form) including Severity and Interference | At each visit up to Week 6 (end of Study)
  Paper questionnaire
Neuropathic Pain Symptom Inventory (NPSI) | Baseline, Week 2, Week 4 and Week 6 (end of Study)
  Paper questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Duan, MD, Study Director — AbbVie
Locations (35):
- United States (19):
  - Site Reference ID/Investigator# 51807, Little Rock, Arkansas
  - Site Reference ID/Investigator# 51946, Anaheim, California
  - Site Reference ID/Investigator# 51468, Long Beach, California
  - Site Reference ID/Investigator# 52744, Walnut Creek, California
  - Site Reference ID/Investigator# 51079, Clearwater, Florida
  - Site Reference ID/Investigator# 51076, Hialeah, Florida
  - Site Reference ID/Investigator# 51945, Hollywood, Florida
  - Site Reference ID/Investigator# 51077, Ocala, Florida
  - Site Reference ID/Investigator# 51078, Orlando, Florida
  - Site Reference ID/Investigator# 51804, Brockton, Massachusetts
  - Site Reference ID/Investigator# 51263, St Louis, Missouri
  - Site Reference ID/Investigator# 51268, St Louis, Missouri
  - Site Reference ID/Investigator# 51302, Omaha, Nebraska
  - Site Reference ID/Investigator# 51271, Flushing, New York
  - Site Reference ID/Investigator# 52743, Portland, Oregon
  - Site Reference ID/Investigator# 51806, Altoona, Pennsylvania
  - Site Reference ID/Investigator# 51265, Tipton, Pennsylvania
  - Site Reference ID/Investigator# 51548, Dallas, Texas
  - Site Reference ID/Investigator# 51269, Renton, Washington
- Czechia (6):
  - Site Reference ID/Investigator# 51425, Hradec Králové
  - Site Reference ID/Investigator# 51426, Mor Ostrava
  - Site Reference ID/Investigator# 51424, Olomouc
  - Site Reference ID/Investigator# 51428, Prague
  - Site Reference ID/Investigator# 51423, Prague
  - Site Reference ID/Investigator# 51427, Zlín
- France (2):
  - Site Reference ID/Investigator# 51924, Le Creusot
  - Site Reference ID/Investigator# 51925, Vénissieux
- Germany (4):
  - Site Reference ID/Investigator# 51503, Berlin
  - Site Reference ID/Investigator# 51642, Düsseldorf
  - Site Reference ID/Investigator# 51502, Mainz
  - Site Reference ID/Investigator# 52346, Münster
- Mexico (4):
  - Site Reference ID/Investigator# 51505, Guadalajara, Jal.
  - Site Reference ID/Investigator# 51504, Mexico City
  - Site Reference ID/Investigator# 51522, Monterrey, N.L.
  - Site Reference ID/Investigator# 51506, Monterrey, N.L.

REFERENCES:
- [Derived] Ziegler D, Duan WR, An G, Thomas JW, Nothaft W. A randomized double-blind, placebo-, and active-controlled study of T-type calcium channel blocker ABT-639 in patients with diabetic peripheral neuropathic pain. Pain. 2015 Oct;156(10):2013-2020. doi: 10.1097/j.pain.0000000000000263. PMID 26067585